CLINICAL TRIAL: NCT00006192
Title: Genetics of Coronary Artery Disease in Alaskan Natives (GOCADAN)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 910; U01HL064244 (NIH)
Record Dates: First submitted 2000-08-31; First posted 2000-09-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Atherosclerosis; Hypertension; Diabetes Mellitus; Coronary Arteriosclerosis
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Atherosclerosis; Hypertension; Diabetes Mellitus; Coronary Artery Disease

SUMMARY:
To document cardiovascular disease and cardiovascular disease risk factors among 1,200 Native Alaskans who are members of approximately 40 families.

DETAILED DESCRIPTION:
BACKGROUND:

There are many compelling reasons to study heart disease in the Native Alaskans. These Eskimo villages are remote and isolated. The traditional lifestyle is being eroded by mechanization and a westernized diet. There has been relatively little outside genetic influence and they are, like the American Indians of the lower 48 states, beginning to show a marked acceleration in the prevalence of atherosclerosis and coronary artery disease.

DESIGN NARRATIVE:

The study is a family-based, cross sectional study. Recognized and emerging risk factors and prevalent cardiovascular disease are documented in each individual through a standardized interview, physical exam, laboratory measurements, carotid ultrasound, ECG, and a review of centralized medical records. Assays will be made of contemporary samples and serum specimens stored at the Anchorage Center CDC antedating this study (10 to 20 years ago) for specific markers of inflammation and serologic responses. Through a ten-centimorgan genetic map, attempts will be made to find specific genes that relate to cardiovascular disease.

The study uses standard methods to assess risk factors relating to lipid metabolism, hypertension, and diabetes mellitus. Importantly, the study also uses state-of-the-art methods for detection of infectious disease exposure, specifically to C. pneumoniae, cytomegalovirus, and other infectious agents hypothesized to play a role in atherogenesis. A case-control age-matched design is used to analyze the infectious disease burden.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Ruotolo — Medstar Health Research Institute

REFERENCES:
- [Background] Nobmann ED, Ponce R, Mattil C, Devereux R, Dyke B, Ebbesson SO, Laston S, MacCluer J, Robbins D, Romenesko T, Ruotolo G, Wenger CR, Howard BV; GOCADAN study, 2000-2003. Dietary intakes vary with age among Eskimo adults of Northwest Alaska in the GOCADAN study, 2000-2003. J Nutr. 2005 Apr;135(4):856-62. doi: 10.1093/jn/135.4.856. PMID 15795447
- [Background] Howard BV, Devereux RB, Cole SA, Davidson M, Dyke B, Ebbesson SO, Epstein SE, Robinson DR, Jarvis B, Kaufman DJ, Laston S, MacCluer JW, Okin PM, Roman MJ, Romenesko T, Ruotolo G, Swenson M, Wenger CR, Williams-Blangero S, Zhu J, Saccheus C, Fabsitz RR, Robbins DC. A genetic and epidemiologic study of cardiovascular disease in Alaska natives (GOCADAN): design and methods. Int J Circumpolar Health. 2005 Jun;64(3):206-21. doi: 10.3402/ijch.v64i3.17985. PMID 16050315
- [Background] Carter EA, MacCluer JW, Dyke B, Howard BV, Devereux RB, Ebbesson SO, Resnick HE. Diabetes mellitus and impaired fasting glucose in Alaska Eskimos: the Genetics of Coronary Artery Disease in Alaska Natives (GOCADAN) study. Diabetologia. 2006 Jan;49(1):29-35. doi: 10.1007/s00125-005-0071-9. Epub 2005 Dec 21. PMID 16369773
- [Derived] Voruganti VS, Cole SA, Ebbesson SO, Goring HH, Haack K, Laston S, Wenger CR, Tejero ME, Devereux RB, Fabsitz RR, MacCluer JW, Umans JG, Howard BV, Comuzzie AG. Genetic variation in APOJ, LPL, and TNFRSF10B affects plasma fatty acid distribution in Alaskan Eskimos. Am J Clin Nutr. 2010 Jun;91(6):1574-83. doi: 10.3945/ajcn.2009.28927. Epub 2010 Apr 21. PMID 20410100